CLINICAL TRIAL: NCT01576627
Title: Zinc Absorption From Zinc Supplements Comparing Zinc Citrate to Zinc Gluconate and Zinc Oxide in Young Adults
Brief Title: Zinc Absorption From Zinc Citrate, Zinc Gluconate and Zinc Oxide
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Michael B. Zimmermann (Other)
Collaborators: University of Zurich (Other)
Responsible Party: Sponsor-Investigator, Prof. Michael B. Zimmermann, Prof, Swiss Federal Institute of Technology
Organization: Swiss Federal Institute of Technology (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: HNL/CTC11-12
Record Dates: First submitted 2012-04-04; First posted 2012-04-12 (Estimated); Last update posted 2013-01-04 (Estimated); Status verified 2013-01

CONDITIONS: Healthy
MeSH Terms: interventions — gluconic acid; Zinc Oxide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- zinc citrate (Experimental)
  Interventions: Dietary Supplement: zinc citrate
- zinc gluconate (Active Comparator)
  Interventions: Dietary Supplement: Zinc Gluconate
- zinc oxide (Active Comparator)
  Interventions: Dietary Supplement: Zinc oxide

INTERVENTIONS:
Dietary Supplement: zinc citrate — 10 mg of zinc as either zinc citrate
  Arms: zinc citrate
Dietary Supplement: Zinc Gluconate — 10 mg of zinc as either zinc gluconate
  Arms: zinc gluconate
Dietary Supplement: Zinc oxide — 10 mg of zinc as either zinc oxide
  Arms: zinc oxide

SUMMARY:
The goal of this trial is to evaluate zinc citrate, a zinc compound with promising sensory properties and a high zinc content, as an alternative zinc compound to be used for supplementation or food fortification. The bioavailability of zinc citrate given as a supplement to young Swiss adults will be assessed and compared to the bioavailability of the commonly used zinc compounds zinc gluconate and zinc oxide.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of 18 to 45 years old
* Body Mass Index in the range of 19 to 25
* No mineral and vitamin supplements two weeks prior to the study and during the whole duration of the study

Exclusion Criteria:

* Any metabolic, gastrointestinal or chronic disease (according to the subjects own statement)
* Long-term medication during the whole study (except for contraceptives)
* Vegans
* Pregnancy
* Lactation
* Intention to become pregnant during the course of the study
* Lack of safe contraception
* Consumption of mineral and vitamin supplements within 2 weeks prior to 1st test supplement administration
* Earlier participation in any nutrition study using Zn stable isotopes as well as participation in any other clinical study within the last 30 days and during this study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2012-03; Primary Completion 2012-05 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Fractional absorption of zinc | 61 days
  Fractional absorption of zinc is estimated by using the double isotope tracer ratio technique by administering 67Zn as oral and 70Zn as intravenous stable isotopes.The urinary enrichment with both isotopes is measured in a spot urine sample by inductively coupled plasma mass spectrometry.

CONTACTS AND LOCATIONS:
Locations (1):
- ETH Zurich, Zurich, Switzerland

REFERENCES:
- [Derived] Wegmuller R, Tay F, Zeder C, Brnic M, Hurrell RF. Zinc absorption by young adults from supplemental zinc citrate is comparable with that from zinc gluconate and higher than from zinc oxide. J Nutr. 2014 Feb;144(2):132-6. doi: 10.3945/jn.113.181487. Epub 2013 Nov 20. PMID 24259556